CLINICAL TRIAL: NCT06847971
Title: Isolated Flexor Hallucis Longus Tendon Transfer VS Gastrocnemius Augmented Flexor Hallucis Longus Tendon Transfer in Management of Achilles Tendon Defect: a Randomized Controlled Trial
Brief Title: Flexor Hallucis Longus Tendon Transfer VS Gastrocnemius Augmented Flexor Hallucis Longus Tendon Transfer in Management of Achilles Tendon Defect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moaiadeldin Ahmed Mohamed Ahmed Abdelmawla, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHLTT VS GAFHLTT in ATD
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Achilles Tendon Repairs/reconstructions; Achilles Tendon Rupture
Keywords: Achilles tendon rupture; flexor hallucis longus; gastrocnemius augmentation; Achilles tendon repairs/reconstructions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flexor hallucis longus tendon transfer (Active Comparator): Achilles tendon defects repair will be done by flexor hallucis longus tendon transfer only.
  Interventions: Procedure: Flexor hallucis longus tendon transfer
- Gastrocnemius augmented flexor hallucis longus tendon transfer (Active Comparator): Achilles tendon defect repair by gastrocnemius augmentation plus flexor hallucis longus tendon transfer
  Interventions: Procedure: Gastrocnemius augmented Flexor hallucis longus tendon transfer

INTERVENTIONS:
Procedure: Flexor hallucis longus tendon transfer — The FHL tendon will be dissected and transected as far distally as possible. The FHL tendon will be transfixed by Krakow's suture being inserted into the distal 3 cm in the stump to ensure adequate length of the graft inserted within the bony tunnel in the calcaneus.A guide wire with eyelet will be inserted in the calcaneum just anterior to the native AT insertion by a distance 2 mm more than the half of the diameter of the transferred tendon to avoid blow up of the posterior wall of the tunnel. A tunnel will be drilled over the guide wire according to the tendon thickness, without penetrating the planter surface of the calcaneum. The threads at the end of FHL tendon suture will be passed through the eyelet of the guide wire. The tendon will be driven into the calcaneal bony tunnel by pulling the guide wire through the plantar aspect of the heel. Then the FHL tendon will be tenodesed into the bone tunnel using a interference screw of the same size or 1 mm larger than the bone tunnel.
  Arms: Flexor hallucis longus tendon transfer
Procedure: Gastrocnemius augmented Flexor hallucis longus tendon transfer — The gastrocnemius tendon will be refixed to the calcaneal tuberosity using anchors. According to the size of the defect: If the size of the gap was 4-5 cm, an additional gastrocnemius turndown or V-Y flaps will be done. Turn down flap will be achieved by creating 2 cm wide and 5-6 cm long flap from the gastrocnemius tendon. The most distal 1 cm from the proximal stump will be secured along the lateral border of the flap to prevent its separation from the original stump during tensioning and fixation to the calcaneus. V-Y flap will be achieved by having inverted V-shaped incision in the distal part of the gastrocnemius starting proximally and extending the two limbs distally leaving the lateral 1 cm from the original tendon. Then carful advancement of the proximal AT stump distally to reach the calcaneal tuberosity. then Fixation will be achieved by suture anchors. If more than 5 cm gap, tenomyodesis of FHL through the proximal stump of Gastrocnemius muscle will be done.
  Arms: Gastrocnemius augmented flexor hallucis longus tendon transfer

SUMMARY:
This study aims to compare the functional outcome of Isolated Flexor hallucis longus tendon transfer and Gastrocnemius Augmented Flexor hallucis longus tendon transfer in repair of Achilles tendon defects. Also, compare the two procedures regarding complication rate, time to restore the function, and the need for secondary procedures.

DETAILED DESCRIPTION:
The Achilles tendon (AT) is the largest and strongest tendon in the human body, yet it is also one of the most commonly ruptured tendons, with an annual incidence of about 18 cases per 100,000 people. Around 75% of Achilles tendon ruptures (ATR) occur in middle-aged patients during sports activity or following trauma. These injuries typically happen in a region 2 to 6 cm above the tendon's attachment to the heel, an area that has a relatively poor blood supply, that reducing the probability of the healing of the tendon by conservative management. Because of the absence of significant pain and the ability to partially maintain plantar flexion, it has been reported that around 10-25% of Achilles tendon rupture (ATR) cases are overlooked or misdiagnosed during the initial medical assessment. The delaying of the diagnosis and by the way the treatment results in a greater separation between the tendon ends, with scar tissue filling the gap leading to lengthening to the gastrocnemius muscle decreasing its tensile forces. This makes the surgical intervention for repair of chronic tendo Achillis rupture necessary to restore normal leg function. Various surgical procedures such as reconstruction with V-Y advanced flap, gastrocnemius turn-down flap, local tendon transfer augments (Flexor hallucis longus (FHL) or peroneus brevis), semitendinosus autograft, free tissue transfer including synthetic grafts and allografts to bridge the gap have been described. Some techniques have been combined, such as tissue advancement and tendon transfer. Multiple studies have been done comparing two or more of the mentioned techniques, but to our knowledge there is no randomized controlled study comparing the isolated FHL tendon transfer to gastrocnemius augmented flexor hallucis longus (GAFHL) tendon transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Adolescents and adults with skeletally mature feet (above 12 y in females and 14 years in males).
* Achilles Tendon defects more than 4 cm resulted from acute or chronic rupture, post-debridement defects in case of neglected insertional tendinopathy, spontaneous ruptures due to tendinosis or after tumor resection.

Exclusion Criteria:

* General medical contraindications to surgical interventions
* Calcaneal Fracture, subtalar fusion
* infection or previous surgery in the ipsilateral hindfoot or ankle
* Systemic disease including seronegative inflammatory diseases, spondyloarthropathies or sarcoidosis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) Score Ankle-Hindfoot Scale | at 6 months, and 1 year follow up visits
  A scale for assessing the functional status of the ankle and hindfoot. It evaluates both subjective and objective components, including pain, function, alignment, and range of motion. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion. Scores range from 0 to 100, and interpreted as: Excellent: 90-100 Good: 80-89 Fair: 70-79 Poor: ≤69
Strength Testing with handheld Dynamometry for plantar flexors | At 3 months, 6 months, and one year follow up visits.
  Isometric plantar flexion against consistent resistance with the strength measured in Newtons.

SECONDARY OUTCOMES:
Rate of complications | Through study completion, an average of 1 year
  wound healing complications, post-operative infections, nerve injuries, and tendon re-rupture.
Foot function index | at 6 months, and 1 year follow up visits
  Foot function index included 17 questions, covering three sub-scales of foot function: Pain, Disability, and Activity Limitation. Scoring for the Foot Function is based on a visual analog scale with 10 intervals. Scores are calculated for each of the sub-scales, as well as a total score (average of all sub-scales). Scores may be represented both as a raw score and a percentage. Higher scores indicate worsening foot health and poorer foot-related quality of life. The score ranges from 0 to 170 with 0 being the best regarding foot function and 170 the worst regarding foot function.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university hospitals, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Guclu B, Basat HC, Yildirim T, Bozduman O, Us AK. Long-term Results of Chronic Achilles Tendon Ruptures Repaired With V-Y Tendon Plasty and Fascia Turndown. Foot Ankle Int. 2016 Jul;37(7):737-42. doi: 10.1177/1071100716642753. Epub 2016 Apr 1. PMID 27036138
- [Background] Nilsson N, Gunnarsson B, Carmont MR, Brorsson A, Karlsson J, Nilsson Helander K. Endoscopically assisted reconstruction of chronic Achilles tendon ruptures and re-ruptures using a semitendinosus autograft is a viable alternative to pre-existing techniques. Knee Surg Sports Traumatol Arthrosc. 2022 Jul;30(7):2477-2484. doi: 10.1007/s00167-022-06943-2. Epub 2022 Apr 9. PMID 35396938
- [Background] Padanilam TG. Chronic Achilles tendon ruptures. Foot Ankle Clin. 2009 Dec;14(4):711-28. doi: 10.1016/j.fcl.2009.08.001. PMID 19857844
- [Background] Gabel S, Manoli A 2nd. Neglected rupture of the Achilles tendon. Foot Ankle Int. 1994 Sep;15(9):512-7. doi: 10.1177/107110079401500912. PMID 7820247
- [Background] Kraeutler MJ, Purcell JM, Hunt KJ. Chronic Achilles Tendon Ruptures. Foot Ankle Int. 2017 Aug;38(8):921-929. doi: 10.1177/1071100717709570. Epub 2017 May 29. No abstract available. PMID 28553729
- [Background] Abraham E, Pankovich AM. Neglected rupture of the Achilles tendon. Treatment by V-Y tendinous flap. J Bone Joint Surg Am. 1975 Mar;57(2):253-5. PMID 1089672
- [Background] Kann JN, Myerson MS. Surgical management of chronic ruptures of the Achilles tendon. Foot and ankle clinics. 1997;2(3):535-45.
- [Background] Cetti R, Junge J, Vyberg M. Spontaneous rupture of the Achilles tendon is preceded by widespread and bilateral tendon damage and ipsilateral inflammation: a clinical and histopathologic study of 60 patients. Acta Orthop Scand. 2003 Feb;74(1):78-84. doi: 10.1080/00016470310013707. PMID 12635798
- [Background] Leslie HD, Edwards WH. Neglected ruptures of the Achilles tendon. Foot Ankle Clin. 2005 Jun;10(2):357-70. doi: 10.1016/j.fcl.2005.01.009. PMID 15922924
- [Background] Abubeih H, Khaled M, Saleh WR, Said GZ. Flexor hallucis longus transfer clinical outcome through a single incision for chronic Achilles tendon rupture. Int Orthop. 2018 Nov;42(11):2699-2704. doi: 10.1007/s00264-018-3976-x. Epub 2018 May 12. PMID 29754186
- [Background] Maffulli N, Waterston SW, Squair J, Reaper J, Douglas AS. Changing incidence of Achilles tendon rupture in Scotland: a 15-year study. Clin J Sport Med. 1999 Jul;9(3):157-60. doi: 10.1097/00042752-199907000-00007. PMID 10512344
- [Background] Leppilahti J, Puranen J, Orava S. Incidence of Achilles tendon rupture. Acta Orthop Scand. 1996 Jun;67(3):277-9. doi: 10.3109/17453679608994688. PMID 8686468